CLINICAL TRIAL: NCT04453410
Title: Validation of a Pediatric Pictorial Version of the QOR-15 Postoperatory Functional Recovery Scale - QoR-15 Pédiatric
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7732
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Surgical Intervention; Minor
Keywords: questionnaire Quality-of-recovery 15 (QoR-15)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire Quality-of-recovery 15 (QoR-15) — Children will use the questionnaire Quality-of-recovery 15 (QoR-15)

SUMMARY:
Consideration from the patient's point of view is an important step in improving postoperative functional recovery. The questionnaire Quality-of-recovery 15 (QoR-15) is a psychometrically validated questionnaire to measure the quality of postoperative functional recovery. it has been recommended in perioperative medecine however, this questionnaire was never adapted and validated for a pediatric surgical population.

The main objective of this protocol is to study the validity, reliability, acceptability and feasibility in routine clinical practice of a pediatric pictorial version of the QoR-15 score.

ELIGIBILITY:
Inclusion Criteria:

* Patient underage over 7 years and up to 17 years and 9 months
* Programming surgery as part of routine management
* Patient affiliated with a health insurance social
* Parental authority holders and the patient agreeing to participate in the study

Exclusion Criteria:

* Patients with severe sensory impairment in preoperation preventing reliable participation in the questionnaire
* Patients at risk of severe cognitive or sensory impairment in postoperative
* Patients with language difficulties in the language of administration of the questionnaire
* Patients who can not express their non-opposition to participation in the study
* Refusal of holders of parental authority and/or refusal of the patient to participate in the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Minor patient over 7 years and up to 17 years and 9 months who have a programming surgery as part of routine management
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Questionnaire Quality-of-recovery 15 score | 3 months
  functional recovery score Questionnaire Quality-of-recovery 15 in pictorial version established at J1 postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Noll E, De Angelis V, Bopp C, Chauvin C, Talon I, Bennett-Guerrero E, Lefebvre F, Pottecher J. Pictorial adaptation of the quality of recovery 15 scale and psychometric validation into a pediatric surgical population. Sci Rep. 2023 Aug 28;13(1):14085. doi: 10.1038/s41598-023-40673-w. PMID 37640781